CLINICAL TRIAL: NCT07093801
Title: Real-world Experience of Lutetium (177Lu) Vipivotide Tetraxetan in Metastatic Castration Resistant Prostate Cancer, an Observational, National, Multicenter, Prospective Cohort Study (PLU4REAL).
Brief Title: Observational Study on Lutetium (177Lu) Vipivotide Tetraxetan to Treat Metastatic Castration Resistant Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAAA617A1IT01
Record Dates: First submitted 2025-07-09; First posted 2025-07-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: Metastatic Castration Resistant Prostate Cancer (mCRPC); lutetium (177Lu) vipivotide tetraxetan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients diagnosed with mCRPC treated with lutetium (177Lu) vipivotide tetraxetan: Adult patients diagnosed with mCRPC eligible for and prescribed with lutetium (177Lu) vipivotide tetraxetan by the treating physician (Multidisciplinary Team).

SUMMARY:
This is a local prospective, multicenter, long-term, non-interventional study using primary data collection to describe the routine clinical practice of patients with mCRPC treated with lutetium (177Lu) vipivotide tetraxetan. The observation period will be from date of start of treatment up to a maximum of 18 months after end of treatment.

ELIGIBILITY:
1. Adult patients diagnosed with mCRPC eligible for and prescribed with lutetium (177Lu) vipivotide tetraxetan by the treating physician (Multidisciplinary Team).
2. ≥ 18 years old at the time of enrollment.
3. Written informed consent must be obtained to participate to this study

In addition to the above-listed criteria, no other inclusion/exclusion criteria exist other than the requirements stated in the local Summary of Product Characteristics (SmPC) and in the "Scheda di Monitoraggio AIFA", e.g., contraindications.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with mCRPC eligible for and prescribed with lutetium (177Lu) vipivotide tetraxetan
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to 18 months post-treatment
  Defined as the time from date of initiation of lutetium (177Lu) vipivotide tetraxetan to the date of first documented progression by investigator assessment (radiographic progression according to the most recent version of Prostate Cancer Working Group [PCWG] or Response Evaluation Criteria In PSMA-PET/CT [RECIP] 1.0, clinical progression, Prostate Specific Antigen [PSA] progression) or death from any cause, whichever occurs first up to 18 months post-treatment.

SECONDARY OUTCOMES:
Second Progression-Free Survival (PFS2) | up to 18 months post-treatment
  Defined as the time from date of initiation of lutetium (177Lu) vipivotide tetraxetan to the date of first documented progression by investigator assessment (radiographic progression according to the most recent version of PCWG or RECIP 1.0, clinical progression, PSA progression) on next-line therapy or death from any cause, whichever occurs first, up to 18 months post-treatment
Overall Survival (OS) | up to 18 months post-treatment
  Defined as the time from of initiation of lutetium (177Lu) vipivotide tetraxetan until death from any cause at each cycle of lutetium (177Lu) vipivotide tetraxetan up to 18 months post-treatment
Prostate-Specific Antigen (PSA) response rates (RR) | up to 18 months post-treatment
  PSA response rates (RR): PSA30; PSA50 and PSA90 while patients are on treatment and up to a maximum of 18 months post-treatment
Overall Response Rate (ORR) | up to 18 months post treatment
  Defined as the proportion of patients with Complete Response (CR) or Partial Response (PR) as Best Overall Response based on RECIST 1.1 or RECIP 1.0.
Duration of Response (DoR) | up to 18 months post-treatment
  Defined as the onset of the first response to disease progression or death for any reason
Proportion of patients with SSE and time to event | up to 18 months post-treatment
  Proportion of patients with Symptomatic Skeletal Event (SSE ) and time to event
Time to initiation of pain medication | from start of treatment to up to 18 months post-treatment
  Time to initiation of pain medication (if not on pain medication at baseline), assessed as time from index date (start of treatment) to date of initiation of pain medication while on treatment or at progression.
Change of pain medication | from baseline to up to 18 months post treatment
  Change of pain medication (dosage or type of medication) at baseline and during treatment/follow-up.
HRQoL - Functional Assessment of Cancer Therapy-Prostate (FACT-P) | from cycle 1 up to 18 months post treatment
  The Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire is a relevant, worldwide tool used for providing insights into both general and prostate-specific concerns in men with prostate cancer.
  The FACT-P is composed of two parts, the FACT-G and the 12-item Prostate Cancer Subscale (PCS). FACT-P total score will be derived as sum of the PWB score, SWB score, EWB score FWB and PCS score and it will range from 0 to 156. Higher scores indicate better health-related quality of life.
HRQoL - Brief Pain Inventory - Short Form (BPI-SF) | from cycle 1 up to 18 months post treatment
  The Brief Pain Inventory - Short Form (BPI-SF) is a widely used tool for assessing clinical pain. The BPI allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function.
  Score ranges from 0 to 10. Higher score indicate worse outcomes.
HRQoL - Functional Assessment of Cancer Therapy - Radionuclide Therapy (FACT-RNT) | from cycle 1 up to 18 months post treatment
  The Functional Assessment of Cancer Therapy - Radionuclide Therapy (FACT-RNT) is used to assess health-related quality of life (HRQoL) in patients undergoing radionuclide therapy for prostate cancer, addressing general concerns and therapy-specific impacts.
  Score ranges from 0 to 60. The higher the score the better the quality of life.
Correlation between baseline clinical and molecular characteristics and and treatment outcomes | from baseline to up to 18 months post treatment
  Correlative analysis between baseline clinical and molecular characteristics (PSA, BRCA 1/2, PET PSMA quantitative analysis and Androgen Receptor [AR] expression) and treatment outcomes (PFS, PFS2, PSA RR, OS, ORR, DOR).
Number of patients with hospitalized infusion of lutetium (177Lu) vipivotide tetraxetan | 8 months (treatment duration period)
  Number of patients with hospitalized infusion of lutetium (177Lu) vipivotide tetraxetan (type of hospitalization and length of stay ).
Number of patients with dosimetry performed | 8-9 months (treatment duration period)
  Number of patients with dosimetry performed before being discharged after infusion of lutetium (177Lu) vipivotide tetraxetan
Number of visits | 9 months (from start of treatment to 30 days FUP period)
  Number of hospitalizations, emergency room visits, and hospital-based outpatient visits between Cycle 1 and the 30-day follow-up period after the last cycle, due to both adverse events (AE) (related or not to the treatment) and events not related to AE
Workdays lost | 8-9 months (treatment duration period)
  Number of workdays lost due to hospitalization for infusion of lutetium (177Lu) vipivotide tetraxetan and number of workdays lost due to hospitalization due to treatment-related AE.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- Italy (23):
  - Novartis Investigative Site, Asti, AT
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Latina, LT
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Rionero in Vulture, PZ
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, La Spezia, SP
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Mestre, VE
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Napoli

IPD SHARING:
Plan to Share IPD: No